CLINICAL TRIAL: NCT02185222
Title: Effect of Vitamin D on Cognitive Decline of Patients With Memory Complaint
Acronym: D-COG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SERC12-TC / D-COG; 2013-005110-36 (EudraCT Number)
Record Dates: First submitted 2014-06-30; First posted 2014-07-09 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Memory Disorders; Age-Related Cognitive Decline
Keywords: Vitamin D; Cholecalciferol; 25-hydroxyvitamin D; Memory complaint; Subjective memory complaint; Mild cognitive impairment; Preventive therapy; Cognitive disorders
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol 100 000 UI (Unité Internationale) (Experimental): Oral solution in single-dose : 100 000 UI per month
  Interventions: Drug: Cholecalciferol 100 000 UI
- Placebo (Placebo Comparator): Oral solution in single-dose per month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol 100 000 UI — Study of superiority between Cholecalciferol high dose 100 000 UI versus placebo : one bulb per month during two years
  Other Names: Uvedose
  Arms: Cholecalciferol 100 000 UI (Unité Internationale)
Drug: Placebo — Study of superiority between Cholecalciferol high dose 100 000 UI versus placebo : one bulb per month during two years
  Arms: Placebo

SUMMARY:
As recommended allowance of oral vitamine D are unable to ensure the recommended serum concentration of vitamine D, the purpose of this study is to show that a dose of vitamin D3 higher than the recommended allowance may slow the cognitive decline of patients with a memory complaint.

ELIGIBILITY:
Pre-Inclusion Criteria :

* Patients aged 60 years or older,
* Who report to a memory centre with symptoms of memory complaint,
* Having a Mini-Mental State Examination (MMSE) score strictly > the 5th percentile for sociocultural level of the patient (GRECO standards for elderly patients),
* Having visual, hearing abilities (authorized equipment) and an oral or written expression sufficient for the suitable realization of the tests,
* Who accept participation in the study and are able to sign the informed consent of the - Affiliated to the French social security system.

Inclusion Criteria:

* Insufficient 25 OH D serum level : 25 OH D < 50 nmol/L (20 ng/ml),
* Normal corrected plasma calcium concentration,
* Normal kidney function (cockcroft > 30 mL/mn)

Exclusion Criteria:

* Alzheimer's disease or other dementia,
* Parkinson's disease treated,
* Epilepsy treated,
* Huntington's disease,
* Brain tumor,
* History of a progressive disease which may have consequences for the central nervous system (blood pressure, higher or equal to 180/100 mmHg, chronic pulmonary disease with hypoxia; cerebrovascular accident of less than 3 months, cranial traumatism with persistent neurologic deficit, subdural hematoma, brain surgery),
* Antecedent of alcoholism or chronic drug-addiction with an obvious or documented consequence on cognition,
* Severe depression : score Montgomery Asberg Depression Rating Scale (MADRS) > 18,
* Psychotropic drug therapy (at the discretion of the clinician),
* Hypercalcaemia or treatment for a hypercalcaemia,
* Known hypersensitivity to the vitamin D,
* Granulomatous disease,
* Treatment of vit D at doses higher than the current recommendations,
* History of calcium urinary lithiasis of less than 1 year,
* Nonsteroidal antiinflammatory drug (NSAID) chronic treatment,
* Severe medical or surgical affection of less than 3 months,
* Unstable health, severe hepatic or renal deficiency,
* Deprivation of liberty, under judicial protection,
* Institutionalization (EHPAD),
* Illiteracy,
* Participation in another biomedical research. A diagnosis of MCI (Mild Cognitive Impairment) of less than 6 months is not a criterion of non-inclusion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline memory functions measured by the score of the total recall test from Free and Cued Selective Recall Reminding Test (Rappel Libre / Rappel Indicé 16 items : RL/RI 16) at one year and at two years | Baseline (at inclusion), one year and two years
  The score of the total recall test from Free and Cued Selective Recall Reminding Test (RL/RI 16) is recommended by a European Task Force consensus.

SECONDARY OUTCOMES:
Changes from baseline global efficiency measured by the Mc Nair scale at one year and at two years | Baseline (inclusion), one year and two years
Evolution of anaemia evaluated by red blood cells count | Baseline (pre-inclusion), one year and two years
Evolution of plasma calcium and albumin concentration | Baseline (pre-inclusion), 45 days, one year and two years
Evolution of urinary calcium and creatinine concentration | 45 days, one year and two years
All adverse events | Up to two years
Serum level of 25-hydroxy vitamine D (25-OH D) measured to study observance | Baseline (pre-inclusion), one year and two years
Changes from baseline global efficiency measured by the Mini Mental State Examination at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline global efficiency measured by the Montreal Cognitive Assessment at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline instrumental activity of daily living measured by 8 items at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline language measured by the "test de denomination orale d'images" (DO-80) at one year and at two years | Baseline (at inclusion), one year and two years
Memory function measured by a visual test : delayed matching to sample 48 items (DMS-48) | Baseline at inclusion
Changes from baseline executive functions measured by the stroop test at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline executive functions measured by the verbal fluency at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline executive functions measured by the Trail Making Test part B at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline attention and speed processing measured by the Trail Making Test part A at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline attention and speed processing measured by the Digit symbol test at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline visuospatial study measured by the Rey figure (copy) at one year and at two years | Baseline (at inclusion), one year and two years
Changes from baseline praxis at one year and at two years | Baseline (at inclusion), one year and two years
  Production of symbolic gesture, imitation utilization gesture, non sense gesture imitation
Changes from baseline depressive symptoms measured by the Montgomery and Asberg Depression Rating Scale at one year and at two years | Baseline (at inclusion), one year and two years

CONTACTS AND LOCATIONS:
Overall Officials: Fanny HENNEKINE, PH, Principal Investigator — CHRU TOURS - Hôpital Bretonneau
Locations (11):
- France (11):
  - Chu Angers, Angers
  - CH BLOIS, Blois
  - CHU BREST - Hôpital de la Cavale Blanche, Brest
  - CHI ELBEUF Louviers Val-de-Reuil, Elbeuf
  - CHU NANTES - Hôpital Bellier, Nantes
  - CHU NANTES - Hôpital Laënnec, Nantes
  - Chr Orleans, Orléans
  - CHU POITIERS - Hôpital de la Milétrie, Poitiers
  - CHU RENNES - Hôpital Hôtel Dieu, Rennes
  - CHU ROUEN - Hôpital Charles Nicolle, Rouen
  - CHRU TOURS - Hôpital Bretonneau, Tours